CLINICAL TRIAL: NCT05837676
Title: Problem-Solving Training for Concussion (PST-Concussion): A Brief, Skills-Focused Intervention to Improve Functional Outcomes in Veterans With mTBI and Co-occurring Mental Health Symptoms
Brief Title: Problem-Solving Training for Concussion
Acronym: PST-Concussion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4778-R; RX004778-01 (Other Grant/Funding Number: VA Rehabilitation Research & Development)
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Brain Concussion
Keywords: Mild Traumatic Brain Injury; Concussion, Mild; Veterans; Neurobehavioral Manifestations; Psychological Distress
MeSH Terms: conditions — Brain Concussion; Neurobehavioral Manifestations | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either PST-Concussion or treatment as usual (TAU).
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors will conduct outcome assessments at 12-week post-test and 24-week follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PST-Concussion (Experimental): Treatment arm. Six, approximately 30-minute telehealth treatment sessions comprised of brief problem-solving training, standard concussion education, motivational interviewing, goal-setting, and compensatory cognitive strategies.
  Interventions: Behavioral: Problem Solving Training for Concussion
- Treatment as usual (TAU) (Other): Control arm. Primary care treatment as usual. Patients assigned to TAU will receive the care that they and their providers determine is necessary to best manage their presenting concerns.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Problem Solving Training for Concussion — PST-Concussion is a combined treatment consisting of brief problem-solving training, standard concussion education, motivational interviewing, goal-setting, and compensatory cognitive strategies.
  Other Names: PST-Concussion
  Arms: PST-Concussion
Other: Treatment as usual — Patients assigned to TAU will receive the care that they and their providers determine is necessary to best manage their presenting concerns.
  Other Names: TAU
  Arms: Treatment as usual (TAU)

SUMMARY:
Mild traumatic brain injury (mTBI), also known as concussion, is a common injury sustained by Veterans. While most individuals who sustain mTBI experience a complete recovery within several weeks of injury, many Veterans with history of mTBI report frequent and long-lasting neurobehavioral complaints and functional impairment. Though research suggests that these outcomes are strongly influenced by co-occurring conditions such as post-traumatic stress disorder, depression, and chronic pain, evidence-based interventions capable of addressing this wide array of concerns are lacking. This study seeks to address this gap by evaluating the effectiveness of a brief and flexible behavioral health treatment (Problem-Solving Training for Concussion, or PST-Concussion), which was designed to be delivered by generalist providers working in VA primary care settings. If PST-Concussion is shown to be effective, this skills-focused intervention may help improve Veterans' recovery experience following mTBI.

DETAILED DESCRIPTION:
This study will be a longitudinal randomized two-arm parallel group clinical trial. Participants will be randomized 1:1 to either PST-Concussion or treatment as usual (TAU). Participants assigned to PST-Concussion will receive six, approximately 30-minute telehealth treatment sessions. Assessments will include standard self-report and cognitive measures that will be administered at baseline, post-treatment, and three-month follow-up. The primary objective of this study will be to evaluate the effectiveness of PST-Concussion in reducing psychological distress compared to TAU. Secondary and tertiary objectives will be to evaluate whether PST-Concussion is associated with appreciable change in subjective neurocognitive functioning, objective neurocognitive functioning, psychosocial functioning, and disability and quality of life. Multi-level modeling will be used to evaluate treatment effects at post-treatment and three-month follow-up. A test of non-inferiority will be conducted to evaluate the potential durability of observed treatment effects from post-test to follow-up. A portion of participants assigned to PST-Concussion will also be interviewed at post-treatment or follow-up to gain insight into the practical impact of intervention on psychosocial functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking Veteran enrolled in VHA care;
* History of concussion (mild traumatic brain injury or mTBI);
* Current psychological distress;
* Subjective neurocognitive symptoms of >= 3 months.

Exclusion Criteria:

* Moderate to severe TBI or other major neurocognitive disorder;
* Psychotic disorder (e.g., schizophrenia spectrum disorder, delusional disorder, bipolar or depressive disorder with psychotic features);
* Acute suicidal ideation;
* Inpatient psychiatric hospitalization within the past 12 months;
* Other illness/ condition that would preclude or predictably influence ability to engage in study visits, as determined by the study team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Brief Symptom Inventory-18 (BSI-18) Global Severity Index T-Score | Up to 24 weeks
  The BSI-18 is a brief measure of psychological distress brought about by common somatic and affective symptoms. It has been validated for use in patients with history of TBI and is appropriate for use in primary care. Similar to a previous trial of PST for mTBI, its Global Severity Index (GSI) T-score will serve as the primary outcome measure. GSI T-scores range from 30-80, with lower scores signaling an overall lower level of psychological distress.

SECONDARY OUTCOMES:
Hopkins Verbal Learning Test-Revised (HVLT-R) | Up to 24 weeks
  A brief test of verbal learning, recall, and recognition. Participants are read a word list over 3 learning trials, and are asked to recall as many words as possible after a 25-minute delay. Raw scores are converted to T-scores (range = <20 to >80), with higher scores signaling better verbal memory performance.
Neurobehavioral Symptom Inventory (NSI) | Up to 24 weeks
  A 22-item checklist of affective, cognitive, and somatosensory symptoms commonly reported after concussion. Scores range from 0 to 88, with lower scores signaling lower overall symptom reports.
Wechsler Adult Intelligence Scale- Fourth Edition (WAIS-IV) Digit Span | Up to 24 weeks
  A brief verbal attention test. Participants are presented with a sequence of digits and asked to repeat them forward and backward. Raw scores are converted to percentile ranks (range = <1 to >99); higher ranks signal better overall performance.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | Up to 24 weeks
  A 26-item abbreviated version of the full-length WHOQOL measure that evaluates disability and quality of life in domains such as social relationships, physical and mental health, and satisfaction with person-environment interactions. Raw scores are averaged to compute domain scores (range = 4-20), with higher scores signaling an overall higher quality of life.
Inventory of Psychosocial Functioning (IPF) | Up to 24 weeks
  An 80-item multidimensional measure of psychosocial functioning and impairment related to mental health symptoms. An overall total is calculated as the mean of all completed subscales, which include: romantic relationships, family, work, friendships and socializing, parenting, education, and self-care. Each domain scale yields a score ranging from 0-100, with higher scores indicating greater impairment.

OTHER OUTCOMES:
Applied Cognition-General Concerns-Short Form (ACGC-8a) | Up to 24 weeks
  An 8-item checklist of general cognitive concerns over the past week. Items were generated and validated as part of the National Institute of Health's Patient-Reported Outcome Measurement Information System (PROMIS). Raw scores are converted to T-scores (range = 23.3-62.7), with higher scores signaling relatively fewer cognitive concerns.
Patient Health Questionnaire-9 (PHQ-9) | Up to 24 weeks
  A 9-item measure of cognitive, affective, and somatic depressive symptoms validated for use in primary care. Scores range from 0 to 27, with lower scores signaling lower mood symptoms.
Applied Cognition-Abilities-Short Form (ACA-8a) | Up to 24 weeks
  An 8-item checklist of self-perceived cognitive abilities over the past week, developed as part of the National Institute of Health's Patient-Reported Outcome Measurement Information System (PROMIS). Raw scores are converted to T-scores (range = 27-64.8) with higher scores signaling higher perceived cognitive abilities.
PTSD Checklist for DSM-5 (PCL5) | Up to 24 weeks
  A 20-item measure of DSM-5 symptoms related to trauma, organized over re-experiencing, avoidance, hyperarousal, and cognitive/mood domains. Score range from 0-80, with lower scores signaling less severe PTSD symptoms.
Alcohol Use Disorders Identification Test (AUDIT) | Up to 24 weeks
  A 10-item measure of the frequency and severity of alcohol intake over the past year. Scores range from 0-40, with higher scores signaling more severe alcohol-related problems.
Pain Symptom Survey (PEG) | Up to 24 weeks
  A 3-item pain assessment that has been validated for use in VA patients. Respondents are asked to report their average level of pain, the average impact of pain on their ability to enjoy life, and the average level of interference on daily activities on a scale of 0 to 10. Ratings on each domain are averaged to calculate a composite score, which ranges from 0 to 10, with lower scores signaling lower overall pain.
Patient Global Impressions of Change (PGIC) | Up to 24 weeks
  A 7-point single-item rating scale that asks patients to rate their overall impression of response to treatment. Ratings range from "no change" to "a great deal better." Ratings range from 0 to 7, with higher ratings signaling greater perceived change in response to treatment.
Community Reintegration of Service-Members (CRIS) | Up to 24 weeks
  A comprehensive measure of community reintegration validated in Veterans with history of mTBI. It consists of 3 subscales that measure extent of participation, satisfaction with participation, and perceived limitations. Individual items are scored on a scale that ranges from 1 to 7, with higher scores signaling more favorable responses.
Drug Abuse Screening Test (DAST10) | Up to 24 weeks
  A 10-item measure of substance misuse and associated functional impairment. Items are rated dichotomously (yes/no), with a total score that ranges from 0 to 10. Higher scores indicate more severe substance use-related problems.
Behavioral Health Measure-20 (BHM-20) | Up to 12 weeks
  A brief measure of emotional distress and life functioning, normed for use in primary care. It consists of 3 subscales that measure general well-being, mental health symptoms, and life functioning. Global mental health scale scores range from 0 to 80, with higher scores signaling greater distress and impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. King, PhD, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY
Locations (1):
- VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the proposed research will be shared outside VA. A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Time Frame: Requests will be considered beginning 6 months after final publication.
Access Criteria: Limited datasets in machine-readable electronic format will be created and shared pursuant to a Data Use Agreement (DUA). Appropriate use of the electronic dataset will be specified, as will prohibitions against identifying or re-identifying (i.e., taking steps to identify or re-identify) any individual whose data are included in the dataset.